CLINICAL TRIAL: NCT00496392
Title: An Open Label, Comparative, Randomised, Balanced Crossover Trial Comparing Nasal Fentanyl and Oral Transmucosal Fentanyl (Actiq®) in Breakthrough Pain in Patients With Cancer
Brief Title: Comparison of Nasal Fentanyl and Oral Transmucosal Fentanyl (Actiq) in Cancer Breakthrough Pain (FT-019-IM)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nycomed (Industry)
Responsible Party: Nycomed, Nycomed
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FT-019-IM; 2006-002087-26
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Pain
Keywords: breakthrough pain in patients with cancer
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Nasal fentanyl — Breakthrough pain in patients with breast or prostate cancer
  Other Names: Instanyl

SUMMARY:
Primary:

• To compare the efficacy of nasal fentanyl (NF) to oral transmucosal fentanyl (Actiq®) (hereafter Actiq) in the management of breakthrough pain in cancer patients.

Secondary:

* To compare patients' general impression and preference of NF and Actiq
* To explore the relationship between NF doses and dose of current opioid for breakthrough pain (BTP) and the relationship between dose of NF and of background opioid
* To assess safety and tolerability of NF

ELIGIBILITY:
Inclusion Criteria:

* Adult in- or out patient with cancer and breakthrough pain; using a stable, chronic opioid treatment for background pain.
* Minimum three BTP episodes per week and maximum four per day. Life expectancy of at least three months.
* Chemotherapy and palliative radiotherapy (except facial radiotherapy) are allowed.
* Randomisation in previous studies with NF, i.e. FT-016-IM, FT-017-IM or FT-018-IM, is not allowed.
* Previous use of Actiq is accepted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2007-01; Primary Completion 2008-08 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Primary endpoint: Time to onset of meaningful pain relief recorded by stopwatch | 26 weeks

SECONDARY OUTCOMES:
• Pain Intensity Differences (PID) at 10 and 30 min derived from Pain Intensity (PI) scores • Sum of Pain Intensity Differences (SPID) 0-15 and 0-60 derived from PI scores • Time to 50% reduction in PI scores • General impression (GI) of the t | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nycomed Clinical Trial Operations, Study Chair — Headquaters
Locations (1):
- Nycomed, Roskilde, Denmark

REFERENCES:
- [Derived] Mercadante S, Radbruch L, Davies A, Poulain P, Sitte T, Perkins P, Colberg T, Camba MA. A comparison of intranasal fentanyl spray with oral transmucosal fentanyl citrate for the treatment of breakthrough cancer pain: an open-label, randomised, crossover trial. Curr Med Res Opin. 2009 Nov;25(11):2805-15. doi: 10.1185/03007990903336135. PMID 19792837